CLINICAL TRIAL: NCT03872479
Title: Open-Label, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Efficacy of EDIT-101 in Adult and Pediatric Participants With Leber Congenital Amaurosis Type 10 (LCA10), With Centrosomal Protein 290 (CEP290)-Related Retinal Degeneration Caused by a Compound Heterozygous or Homozygous Mutation Involving c.2991+1655A>G in Intron 26 (IVS26) of the CEP290 Gene ("LCA10-IVS26")
Brief Title: Single Ascending Dose Study in Participants With LCA10
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Editas Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1991-201-008
Record Dates: First submitted 2018-10-12; First posted 2019-03-13 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Leber Congenital Amaurosis 10; Inherited Retinal Dystrophies; Eye Diseases, Hereditary; Retinal Disease; Retinal Degeneration; Vision Disorders; Eye Disorders Congenital
Keywords: CEP290; LCA10; Retinal degenerative diseases (RDD); Leber congenital amaurosis (LCA); Congenital Retinal Blindness; p.Cys998X; c.2991+1655A>G; CRISPR Treatment; Cas9 Protein; Eye Diseases Signs and Symptoms; Genetic Diseases, Inborn; Congenital Abnormalities; Eye Abnormalities; CRISPR-Cas9; CRISPR Associated Protein 9; Cas9 Enzyme
MeSH Terms: conditions — Leber Congenital Amaurosis 10; Eye Diseases, Hereditary; Retinal Diseases; Retinal Degeneration; Vision Disorders; Eye Abnormalities; Meckel Syndrome, Type 4; Leber Congenital Amaurosis; Genetic Diseases, Inborn; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Adults Low Dose (Experimental): Single dose of EDIT-101 administered by subretinal injection surgery
  Interventions: Drug: EDIT-101
- Adults Middle Dose (Experimental): Single dose of EDIT-101 administered by subretinal injection surgery
  Interventions: Drug: EDIT-101
- Adults High Dose (Experimental): Single dose of EDIT-101 administered by subretinal injection surgery
  Interventions: Drug: EDIT-101
- Pediatric Middle Dose (Experimental): Single dose of EDIT-101 administered by subretinal injection surgery
  Interventions: Drug: EDIT-101
- Pediatric High Dose (Experimental): Single dose of EDIT-101 administered by subretinal injection surgery
  Interventions: Drug: EDIT-101

INTERVENTIONS:
Drug: EDIT-101 — Participants will receive a single dose of EDIT-101 administered via subretinal injection in the study eye. Up to 5 cohorts across 3 doses will be enrolled in this study.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of a single escalating doses of EDIT-101 administered via subretinal injection in participants with LCA10 caused by a homozygous or compound heterozygous mutation involving c.2991+1655A>G in intron 26 of the CEP290 gene ("LCA10-IVS26").

DETAILED DESCRIPTION:
This is an open-label, single ascending dose study of EDIT-101 in adult and pediatric (ie, ages 3 to 17) participants with LCA10-IVS26. Up to 34 participants will be enrolled in up to 5 cohorts to evaluate up to 3 dose levels of EDIT-101 in this study. EDIT-101 is a novel gene editing product designed to eliminate the mutation on the CEP290 gene that results in the retinal degeneration that defines LCA10-IVS26.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least 3 years of age at screening with CEP290-related retinal degeneration caused by a homozygous or compound heterozygous mutation involving c.2991+1655A>G in IVS26 of the CEP290 gene.
* Visual Acuity:

  * Sentinel participant will have severe vision loss with a logMAR BCVA of ≥1.6 to 3.9 (20/800 or worse to LP) in the study eye
  * Non-sentinel participants must have BCVA between 1.0 - 3.0 logMAR in the study eye

Exclusion Criteria:

* Other known disease-causing mutations
* Achieves a passing score for the mobility course at the most difficult level
* In either eye, active systemic or ocular/intraocular infection or inflammation
* In either eye, history of steroid-responsive intraocular pressure with increases > 25 mm Hg following corticosteroid exposure
* Any vaccination/immunization in the last 28 days before screening
* Inability or unwillingness to take oral prednisone
* Prior gene therapy or oligonucleotide treatment

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-05-23 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events related to EDIT-101 | 1 year
Number of participants experiencing procedural related adverse events | 1 year
Incidence of dose limiting toxicities | 1 year

SECONDARY OUTCOMES:
Maximum tolerated dose as determined by occurrence of dose limiting toxicities | 1 year
Change from baseline in Mobility course score | 1 year
  Testing the subjects visual function by having the subject walk through obstacle courses. Courses will have different levels of difficulty depending on the light levels of the room and the contrast of the objects in the room.
Change from baseline in LogMAR measurement of BCVA | 1 year
  The test will evaluate visual acuity in ranges from light perception to normal vision.
Change from baseline in pupillary response | 1 year
  Measuring the change in pupil diameter in response to a light stimulus.
Change from baseline in dark adapted visual sensitivity using Full field light sensitivity threshold (FST) | 1 year
  Flashes of light of varying luminance are presented to the eye and the subject reports is the flash was seen.
Change from baseline in macula thickness | 1 year
Change from baseline in contrast sensitivity | 1 year
  The Lea symbols chart will be used for subjects under age 6 and the Pelli-Robson chart for all other subjects. The images or letters on the charts are in decreasing contrast.
Change from baseline in macular sensitivity as measured by microperimetry | 1 year
  Visual field test measuring the amount of light perceived in specific parts of the macula.
Change from baseline in color vision score using the Farnsworth 15 score | 1 year
  The Farnsworth D15 tests for congenital and acquired color vision defects. Fifteen color discs will be arranged by the subject. Scoring is accomplished by recording the sequence selected by the patient on a copy of the score sheet. A patient with a color vision deficiency will arrange the color discs in a different order than a person with normal color vision.
Change from baseline in QOL score for Age <8 years using the Children's Visual Function Questionnaire | 1 year
Change from baseline in QOL score for Age 8 to <18 years using the Impact of Vision Impairment for Children | 1 year
Change from baseline in QOL score for Age >18 years if BCVA is worse than 1.0 logMAR in both eyes using the Impact of Vision Impairment for Very Low Vision | 1 year
Change from baseline in QOL score for Age >18 years if BCVA is 1.0 logMAR or better in both eyes using the Impact of Vision Impairment | 1 year
Change from baseline in visual field using kinetic perimetry | 1 year
  Kinetic perimetry looks as the visual field to identify regions of normal and abnormal sensitivity to light
Change from baseline in Patient Global Impressions of Change score | 1 year
  This QOL has 5 non-numeric choices for the subject to select how they believe their condition has changed.
Change from baseline in gaze tracking | 1 year
  Video clips of the eyes are used to measure eye position and stability over time.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Bascom Palmer Eye Institute, Miami, Florida
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - W.K. Kellogg Eye Center - University of Michigan, Ann Arbor, Michigan
  - Casey Eye Institute - OSHU, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pierce EA, Aleman TS, Jayasundera KT, Ashimatey BS, Kim K, Rashid A, Jaskolka MC, Myers RL, Lam BL, Bailey ST, Comander JI, Lauer AK, Maguire AM, Pennesi ME. Gene Editing for CEP290-Associated Retinal Degeneration. N Engl J Med. 2024 Jun 6;390(21):1972-1984. doi: 10.1056/NEJMoa2309915. Epub 2024 May 6. PMID 38709228
- [Derived] Harvey JP, Sladen PE, Yu-Wai-Man P, Cheetham ME. Induced Pluripotent Stem Cells for Inherited Optic Neuropathies-Disease Modeling and Therapeutic Development. J Neuroophthalmol. 2022 Mar 1;42(1):35-44. doi: 10.1097/WNO.0000000000001375. Epub 2021 Sep 30. PMID 34629400
- [Derived] Zhang X, Zhang D, Thompson JA, Chen SC, Huang Z, Jennings L, McLaren TL, Lamey TM, De Roach JN, Chen FK, McLenachan S. Gene correction of the CLN3 c.175G>A variant in patient-derived induced pluripotent stem cells prevents pathological changes in retinal organoids. Mol Genet Genomic Med. 2021 Mar;9(3):e1601. doi: 10.1002/mgg3.1601. Epub 2021 Jan 26. PMID 33497524